CLINICAL TRIAL: NCT05265234
Title: Monitoring Response to Therapy in Atopic Dermatitis Patients Treated With Dupilumab Using Noninvasive Reflectance Confocal Microscopy and Optical Coherence Tomography
Brief Title: Dupilmuab for Atopic Dermatitis Monitored With Noninvasive Imaging.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OptiSkin Medical (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Orit Markowitz MD, Medical Director, OptiSkin Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTI-003
Record Dates: First submitted 2021-12-16; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: dermatitis; Dupilumab; Inflammatory Skin Diseases; itch relief; biologic
MeSH Terms: conditions — Eczema; Dermatitis, Atopic; Dermatitis | interventions — dupilumab; Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dupixent (Experimental): Patients will receive initial dose of 600 mg (two 300 mg injections in different injection sites), followed by 300 mg given every other week for 16 weeks.
  Patients will self-administer by subcutaneous injection at home, instructions will be provided at first visit.
  Interventions: Drug: Dupilumab; Device: Optical Coherence Tomography; Device: Reflectance confocal microscopy

INTERVENTIONS:
Drug: Dupilumab — IL-4 antagonist to improve moderate-severe atopic dermatitis
  Other Names: Dupixent
Device: Optical Coherence Tomography — OCT is a noninvasive imaging device that can be used to monitor inflammatory skin disorders.
  Other Names: OCT
Device: Reflectance confocal microscopy — RCM is a noninvasive imaging device, with resolution approaching that of histology, which can monitor structural changes in the epidermis and superficial dermis, monitor inflammatory cells, and can overcome the limitations of a traditional biopsy.
  Other Names: RCM

SUMMARY:
The study is trying to answer the following question: "Can we use non-invasive imaging to evaluate the response of atopic dermatitis (eczema) to Dupixent (dupilumab)?"

DETAILED DESCRIPTION:
Participating in this research will allow the subject to undergo a noninvasive imaging alternative to conventional monitoring in response to a biologic. Normally, subjects would undergo a clinical examination, serial photography, and possible biopsies to assess the progression of the disease. This study will get rid of the need for a biopsy but will require multiple scans with non-invasive imaging. This research examines a new approach to monitoring response to a biologic drug used for atopic dermatitis, and can also, be used to grade disease severity without the need for a biopsy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Atopic dermatitis (AD) affecting ≥10% body surface area (BSA) at baseline
* IGA score ≥3, on the IGA scale of 0-4 at baseline
* Eczema Area and Severity Index (EASI) score of ≥16 at baseline

Exclusion Criteria:

* Prior treatment with Dupilumab (REGN668/SAR231893)
* Treatment with TCS or topical calcineurin inhibitors (TCI) within 2 weeks before the baseline visit
* Bodyweight <30 kg (65lb) at Baseline
* Known or suspected immunodeficiency including human immunodeficiency virus (HIV) infection
* Pregnancy, breastfeeding or planning to become pregnant or breastfeed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Baseline to 16 weeks
  The Eczema Area and Severity Index (EASI) is a tool used to measure the extent (area) and severity of atopic eczema, ranging 0-72, 0 being least severe and 72 being most severe.
Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) | Baseline to 16 weeks
  Investigator will use the Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) a tool used to measure the severity of atopic eczema, ranging 0-4, 0 is clear and 4 is most severe.
Noninvasive Imaging (clinical response) with Reflectance Confocal Microscopy (RCM) | Baseline to 16 weeks
  Reflectance Confocal Microscopy (RCM) is a noninvasive imaging device that can be used to monitor the severity of inflammatory skin disorders without the need for a biopsy. RCM can visualize cells with a resolution comparable to a light microscope, allowing the investigators to identify the degree of inflammation and damage to the skin.
  An overall disease severity score ranging from 0-3 (0=none, 1=mild, 2= moderate, 3=severe) will use aggregates of the following *features:
  * Spongiosis
  * Parakeratosis
  * Epidermal thickness
  * Quality of honeycomb structure of the stratum spinosum
  * Appearance of the dermal-epidermal junction
  * Appearance of the superficial dermis
  * Recognition of the dermal papilla
  * Caliber of blood vessels
  * Presence of inflammatory cells
    * Grading will be scored (0=none, 1=mild, 2= moderate, 3=severe), a greater numerical score indicates more advanced disease.
Noninvasive Imaging (clinical response) with Optical Coherence Tomography (OCT) | Baseline to 16 weeks
  Optical Coherence Tomography (OCT) is a noninvasive imaging device that can be used to monitor the severity of inflammatory skin disorders without the need for a biopsy. OCT can detect deep structures in the skin, identify areas of inflammation, and determine the thickness of the skin. These measures will be consolidated to a severity score ranging 0-3, (0= no disease, 3= severe disease) and will be tracked throughout the duration of the study.
  The following features will be aggregated to form an Optical Coherence Tomography-severity-score:
  * Change in the epidermal thickness
  * Changes in anatomy or appearance of the dermo-epidermal junction and the dermis.
  * Changes in vascular flow patterns, including the number and density of vessels in skin using the dynamic feature of Optical Coherence Tomography
    * Grading will be scored 0=none, 1=mild, 2= moderate, 3=severe

CONTACTS AND LOCATIONS:
Overall Officials: Orit Markowitz, MD, Principal Investigator — Medical Director
Locations (1):
- OptiSkin Medical, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leung DY, Guttman-Yassky E. Deciphering the complexities of atopic dermatitis: shifting paradigms in treatment approaches. J Allergy Clin Immunol. 2014 Oct;134(4):769-79. doi: 10.1016/j.jaci.2014.08.008. PMID 25282559
- [Background] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Background] Meinke MC, Richter H, Kleemann A, Lademann J, Tscherch K, Rohn S, Schempp CM. Characterization of atopic skin and the effect of a hyperforin-rich cream by laser scanning microscopy. J Biomed Opt. 2015 May;20(5):051013. doi: 10.1117/1.JBO.20.5.051013. PMID 25467783
- [Background] Byers RA, Maiti R, Danby SG, Pang EJ, Mitchell B, Carre MJ, Lewis R, Cork MJ, Matcher SJ. Sub-clinical assessment of atopic dermatitis severity using angiographic optical coherence tomography. Biomed Opt Express. 2018 Mar 29;9(4):2001-2017. doi: 10.1364/BOE.9.002001. eCollection 2018 Apr 1. PMID 29675335
- [Background] Tang TS, Bieber T, Williams HC. Are the concepts of induction of remission and treatment of subclinical inflammation in atopic dermatitis clinically useful? J Allergy Clin Immunol. 2014 Jun;133(6):1615-25.e1. doi: 10.1016/j.jaci.2013.12.1079. Epub 2014 Mar 18. PMID 24655575
- See also: FDA Approved Drugs: Dupixent — https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=BasicSearch.process